CLINICAL TRIAL: NCT04043117
Title: Body Image and Self-esteem in a Sample of Oncological Adolescents: A Pilot Study
Brief Title: Body Image and Self-esteem in Adolescence
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to covid-19 sanitary restrinction in the oncology ward and day hospital.
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: Dimorphism and Self-esteem
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-10

CONDITIONS: Body Image
Keywords: Dimorphism; self-esteem; oncological treatments

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clinical Group: Group is composed by 12-19 years adolescents with a tumor (excluding brain tumor). Every patient included in the group complete the assessment including: evaluation of self-esteem (TMA test) and body image (BUT test, I-BICI test and Human Figure Drawing).
  Interventions: Other: Body Image evaluation; Other: Self esteem evaluation

INTERVENTIONS:
Other: Body Image evaluation — Evaluation of body image perception requires three assessment tools administered at four different times:
  T0: During the first week of admission T1: Three months from the first admission T2: Six months from the first admission T3: One year from the end of the treatment
  1. Italian Body Image Concern Inventory: 19-items self-report instrument rated on a 5-points Likert scale (1 = never; 5 = always). It consists of two sub-scales to evaluate body image-related dissatisfaction and concern respectively.
  2. Body Uneasiness Test: 71-item self-report questionnaire on a 6-points Likert scale (0 = never; 5 = always) that consists of two subscales: BUT-A (measuring weight phobia, body image concerns, avoidance, compulsive self-monitoring, detachment and body depersonalization) and BUT-B (measuring worries about specific body parts or functions).
  3. Human Figure Drawing: qualitative measure of adolescent's body perception; participants are asked a free draw, representing themselves.
Other: Self esteem evaluation — Evaluation of body image perception is achieved administering TMA test at four different times:
  T0: During the first week of admission T1: Three months from the first admission T2: Six months from the first admission T3: One year from the end of the treatment
  TMA (Multidimensional Self-Esteem Test): a 150-items self-report questionnaire for children and adolescents from 9 to 19 years old. It's made up of six subscales: interpersonal relationships, environmental control competence, emotionality, scholastic success, family life, body perception. Participants have to express their agreement with each item according to the following response options: absolutely true, true, false, absolutely false.

SUMMARY:
To evaluate the difference between body image and self-esteem scores during and at the end of the medical. Hypothesis: body image and self-esteem changes during the oncological treatments.

DETAILED DESCRIPTION:
Body image and self-esteem represent important variables linked to adolescents' development. These two variables are the most affected in patients with the oncological disease.

The consequences of a visible difference may have a significant impact on behaviour and mood, causing relevant impairments in individuals well-being and quality of life. Among different personal attributes, self-esteem may be the one with the greatest impact on body image (Cash, 2002). Indeed previous studies have investigated different features of body image and self-esteem (Webster & Tiggemann, 2003), showing that they have a significant influence on the overall well-being (Cash & Fleming, 2002), and that those aspects are also significantly influenced by age and gender. The patients are evaluated at T0 (within the first week of hospitalization after diagnosis), T1 (within 3 months after diagnosis), T2 (within 6 months after diagnosis), T3 (within 12 months after diagnosis, at the end of cancer treatment), according to a follow-up study design. Data analysis: r Pearson's correlation, repeated measure ANOVA and regression analysis will be carried out to investigate relations between studied variables and eventual changes over time. Analyses are performed using SPSS software (Chicago, S. P. S. S. SPSS Inc; 2008. SPSS Statistics, 17.)

ELIGIBILITY:
Inclusion criteria for patients:

* Age between 12 and 19 years
* Adequate knowledge of the Italian language
* Consent to participation
* First diagnosis for oncological pathology of leukaemia or bone cancer

Exclusion criteria for pediatric patients:

* Patients under the age of 12 or over 19 years
* Not adequate knowledge of the Italian language
* Patients who have a relapse with respect to the pathology already treated
* Patients with previous oncological diseases
* Cognitive disability
* Patients with brain tumours
* Patients with gender dysphoria
* Absence of informed consent
* Previous diagnosis of Anxiety or Depression
* Diagnosis of an eating disorder

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Adolescents considered suitable to participate in the study on the basis of the inclusion criteria will be recruited by the investigator in the Oncohematology department and Day Hospital of the same department during the first hospitalization following the communication of the diagnosis
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Image perception during the path of illness | Evaluation at T0 (within the first week of hospitalization after diagnosis), T1 (within 3 months after diagnosis), T2 (within 6 months after diagnosis), T3 (within 12 months after diagnosis, at the end of cancer treatment).
  I-BICI (Italian Body Image Concern Inventory): a self-report instrument composed by 19 items rated on a 5-points Likert scale (1 = never; 5 = always). It consists of two sub-scales to evaluate body image-related dissatisfaction and concern respectively. BUT (Body Uneasiness Test): a 71-item self-report questionnaire on a 6-points Likert scale (0 = never; 5 = always) that consists of two subscales: BUT-A which measures weight phobia, body image concerns, avoidance, compulsive self-monitoring, detachment and estrangement feelings towards one's own body (depersonalization); and BUT-B, which looks at specific worries about particular body parts or functions.
Change in self esteem levels during the path of illness | Evaluation at T0 (within the first week of hospitalization after diagnosis), T1 (within 3 months after diagnosis), T2 (within 6 months after diagnosis), T3 (within 12 months after diagnosis, at the end of cancer treatment), according to a foll
  TMA (Multidimensional Self-Esteem Test): a 150-items self-report questionnaire for children and adolescents from 9 to 19 years old. It's made up of six subscales: interpersonal relationships, environmental control competence, emotionality, scholastic success, family life, body perception. Participants have to express their agreement with each item according to the following response options: absolutely true, true, false, absolutely false

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Martin, MSc, Principal Investigator — Head of Pediatric Psychology
Locations (1):
- Meyer Children's Hospital, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision has to be shared with the local Clinical Trial Office of the Hospital

REFERENCES:
- [Background] Cash TF, Fleming EC. The impact of body image experiences: development of the body image quality of life inventory. Int J Eat Disord. 2002 May;31(4):455-60. doi: 10.1002/eat.10033. PMID 11948650
- [Background] Gatti, E., Ionio, C., Traficante, D., & Confalonieri, E. (2014). "I Like My Body; Therefore, I Like Myself": How Body Image Influences Self-Esteem-A Cross-Sectional Study on Italian Adolescents. Europe's Journal of Psychology, 10(2), 301-317.
- [Background] Pendley JS, Dahlquist LM, Dreyer Z. Body image and psychosocial adjustment in adolescent cancer survivors. J Pediatr Psychol. 1997 Feb;22(1):29-43. doi: 10.1093/jpepsy/22.1.29. PMID 9019046
- [Background] Armstrong-James L, Cadogan J, Williamson H, Rumsey N, Harcourt D. An evaluation of the impact of a burn camp on children and young people's concerns about social situations, satisfaction with appearance and behaviour. Scars Burn Heal. 2018 Dec 10;4:2059513118816219. doi: 10.1177/2059513118816219. eCollection 2018 Jan-Dec. PMID 30574405
- [Background] Stormer SM, Thompson JK. Explanations of body image disturbance: a test of maturational status, negative verbal commentary, social comparison, and sociocultural hypotheses. Int J Eat Disord. 1996 Mar;19(2):193-202. doi: 10.1002/(SICI)1098-108X(199603)19:23.0.CO;2-W. PMID 8932558
- [Background] Webster J, Tiggemann M. The relationship between women's body satisfaction and self-image across the life span: the role of cognitive control. J Genet Psychol. 2003 Jun;164(2):241-52. doi: 10.1080/00221320309597980. PMID 12856818
- [Background] Wardle J, Beales S. Restraint, body image and food attitudes in children from 12 to 18 years. Appetite. 1986 Sep;7(3):209-17. doi: 10.1016/s0195-6663(86)80026-5. PMID 3800362